CLINICAL TRIAL: NCT05223114
Title: Airway Microbiome and Th17-mediated Inflammation in COPD Among HIV-infected Individuals in a Rural Ugandan Cohort
Acronym: HLM
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: MHREC2152; TMA2020CDF-3194 (Other Grant/Funding Number: EDCTP)
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: COPD; HIV Infections; Respiratory Disease
Keywords: airway microbiome; COPD; HIV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; HIV Infections; Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Induced sputum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV+COPD+: 40 male and female adults > 35 years with COPD and HIV
  Interventions: Other: Not applicable (N/A)
- HIV+COPD-: 40 male and female adults > 35 years with HIV but no COPD
  Interventions: Other: Not applicable (N/A)
- HIV-COPD+: 40 male and female adults > 35 years with COPD not HIV
  Interventions: Other: Not applicable (N/A)
- HIV-COPD-: 40 male and female adults > 35 years with no COPD and no HIV
  Interventions: Other: Not applicable (N/A)

INTERVENTIONS:
Other: Not applicable (N/A) — Not applicable to this study

SUMMARY:
Rationale: COPD is increasing in prevalence among people living with HIV/AIDS (PLWHA) as widespread use of ART has increased longevity in this population. In rural Ugandan ART clinics, we report COPD prevalence of 6.22%. Currently, it's not fully known what drives chronic lung inflammation in PLWHA population despite being virologically suppressed on ART. There is need to explore factors driving chronic airway inflammation among PLWHA. Airway microbiome has been implicated in the pathogenesis of COPD. Preliminary analysis from our study revealed that, specific microbes were significantly enriched in PLWHA with COPD with more lung bacteria impacted by HIV than COPD. These findings suggest that HIV-associated changes in unique airway microbial genera may be driving COPD among PLWHA in our cohort. Currently, we don't know how such genera drive chronic airway inflammation.

Study objectives: In this study, we will: (1) establish a relationship between airway microbiome and Th17/Treg cellular phenotypes among HIV-infected individuals with COPD; (2) investigate bacterial-mediated Th17 upregulation of pro-inflammatory and pro-fibrotic genes among HIV individuals with COPD and (3) explore the role of bacterial outer membrane vesicles (OMVs) in mediating microbiome driven Th17 immune responses among HIV individuals.

Methods: We will conduct a 2-year case-controlled study, leveraging on the established lung microbiome cohort in rural Nakaseke district of Uganda. We will recruit 80 HIV-infected individuals ≥35 years attending the ART clinic at Nakaseke General Hospital screened for COPD as well as 80 HIV-negative controls ≥35 years attending the pulmonary clinic at Nakaseke General Hospital screened for COPD. In both cases and controls, we will consider 40 stable COPD participants and 40 participants with no COPD. Recruited participants will undergo sputum induction protocol at our newly established negative pressure sputum induction facility at Nakaseke General Hospital following established standard operating procedures. Using induced sputum samples, we will (i) perform 16S sequencing and metagenomics analysis to determine airway bacterial communities, (ii) RNA sequencing and analysis to determine gene expression profiles, mass flow cytometry and analysis to profile immune cells in induced sputum of study participants as well as (iv) ELISA tests to compare OMV levels between participants.

DETAILED DESCRIPTION:
Introduction The improvement in access to antiretroviral therapy (ART) among people living with HIV/AIDs (PLWHA) has resulted in a decrease in HIV-associated morbidity and mortality[1]. This is particularly true in low- and middle-income countries (LMICs), which bear the largest burden of HIV[2]. The reduction in mortality has substantially increased life expectancy, with estimates among PLWHA now approaching that of the general population[3]. Consequently, there has been increased attention among survivors to the emerging burden of non-communicable diseases (NCD), such as chronic obstructive pulmonary disease (COPD)[4]. Sub-Saharan Africa, which has the highest density of PLWHA, has experienced dramatic increases in COPD related-morbidity and mortality especially in individuals with history of pulmonary tuberculosis (PTB)[5]. In rural Ugandan ART clinics, we reported COPD prevalence of 6.22% with history of PTB being the strongest predictor of COPD risk and reduced lung function[5]. Currently, it's not fully known what drives chronic lung inflammation in PLWHA population well-controlled on ART.

In search for answers to the above question, we have been exploring the role of altered airway microbiome in orchestrating chronic airway inflammation in PLWHA. Our research question has been supported by a growing body of knowledge from human and animal studies that alterations in the bacterial communities inhabiting the airway trigger immune responses and chronic airway inflammation[6-9]. In a recent study involving 50 HIV+COPD+, 50 HIV+COPD-, 50 HIV-COPD- and 50 HIV-COPD- participants in rural Uganda, we investigated the association between altered airway microbiome and HIV-associated COPD (NCT040702). Preliminary analysis from 16S sequencing on induced sputum samples revealed that, in spite of minor differences in bacterial diversity among PLHWA with COPD compared to controls, commensal microbes belonging to the genera Atopobium, Megasphaera, Actinomyces, Selenomonas, Stomatobaculum and Oribacterium were significantly enriched in PLWHA with COPD while microbes belonging to the genera Prevotella, Porphyromonas, Pseudopropionibacterium, Odoribacter and Filifactor were depleted. Our results clearly show that there are more lung bacteria impacted by HIV than COPD, suggesting that HIV-associated changes in unique airway microbial genera may be driving COPD among PLWHA in our cohort. Currently, what remains unknown is how such genera drive chronic airway inflammation.

Studies from mouse models report Prevotella, Bacteroides and Veillonella to play a significant role in orchestrating lung inflammation through Toll like receptor (TLR) 2/4 signaling on alveolar macrophages, epithelial cells and dendritic cells which prime cells of the adaptive immunity[8]. The reported outcome has been aberrant Th17 and reduced Treg immune responses using germ-free and specific pathogen-free mice models [8]. Similarly, recent evidence in human studies show that Prevotella and Veillonella genera are associated with a distinct metabolic profile, enhanced pro-inflammatory cytokine expression characterized by elevated Th17 cellular response[9]. Microbiome-host cell communication has been reported to be mediated by secreted bacterial outer membrane vesicles (OMVs), which correlate with bacterial biomass (figure 2) [8]. We believe that identifying airway bacterial genera which elicit aberrant Th17 response among PLWHA with COPD could be a stepping stone towards developing strategies aimed at restoring microbial balance either through direct elimination of pathobionts by antibiotics or restoration of commensals through probiotics to promote colonization resistance at mucosal surfaces.

Based on this background, we aim to investigate if airway microbiome fuels Th17 mediated airway inflammation in COPD among HIV-infected individuals. We hypothesize that: (1) microbiome induces airway Th17 and suppresses Treg immune responses among HIV-infected individuals with COPD; (2) bacterial-driven Th17 response promotes expression of pro-inflammatory genes among individuals with COPD and (3)airway microbiome mediates its effect on Th17 immune response through secretion of bacterial outer membrane vesicles (OMVs).

In this study, we will: (1) establish a relationship between airway microbiome and Th17/Treg cellular phenotypes among HIV-infected individuals with COPD; (2) investigate bacterial-mediated Th17 upregulation of pro-inflammatory and pro-fibrotic genes among HIV individuals with COPD and (3) explore the role of bacterial outer membrane vesicles (OMVs) in mediating microbiome driven Th17 immune responses among HIV individuals.

Study aims and objectives

Study aim:

To investigate airway microbiome-driven Th17 mediated inflammation in COPD among HIV-infected individuals

Specific objectives

1. To establish a relationship between airway microbiome and Th17/Treg cellular phenotypes among HIV-infected individuals with COPD.
2. To investigate bacterial mediated Th17 upregulation of pro-inflammatory genes among HIV-infected individuals with COPD
3. To investigate the role of bacterial outer membrane vesicles (OMVs) in mediating dysbiosis driven Th17 immune responses among HIV individuals.

Problem statement Chronic obstructive pulmonary disease is increasing in prevalence among people living with HIV/AIDS (PLWHA) as widespread use of Antiretroviral Therapy (ART) has increased longevity in this population[5]. It is still unknown what drives chronic airway inflammation in PLWHA well controlled on ART. In spite of a well-established association between COPD and pulmonary tuberculosis, it does not fully account for the reported cases of COPD among PLWHA[5]. In our study population, neither smoking nor biomass exposure have been reported to be associated with COPD. There is need to explore factors driving chronic airway inflammation among PLWHA.

Justification Specific microbial communities capable of eliciting intense immune responses could determine the outcome of host-microbiome interaction, being either immune tolerance or inflammation. Whereas in-depth characterization of airway microbiome has been performed in COPD human studies and animal models[5-8], only associations have been reported and a few specific signatures have been implicated as predictors of COPD mortality[9]. Few animal-based, microbiome models have been translated into testable human airway or lung-based model to elaborate on the mechanistic role of microbiome in COPD. Deciphering which bacteria induce a strong immune response amidst a multitude of microbial communities remains a significant area of interest to sub phenotype and identify treatable traits. We believe that pursuit of this research question will provide a basis for immunophenotyping airway microbial communities as tolerogenic (Treg-inducing) or inflammatory (Th17-inducing), a potentially seminal scientific discovery in respiratory immunobiology.

Literature review Globally more than 80% of NCD-related deaths occur in Low-and-Middle-Income Countries (LMIC)[10]. Among NCDs, chronic lung disease is the fourth leading cause of death worldwide and is predicted to be the third-largest health problem in Sub-Saharan Africa by 2030[11]. COPD is a progressive life-threatening airflow obstruction that causes breathlessness initially with exertion and predisposes to exacerbations and serious illness[12]. In the general population, COPD had claimed a total of three million lives globally by 2015[13]. As a result of the global scale-up of antiretroviral therapy (ART) and cotrimoxazole prophylaxis, the incidence of pulmonary infections has declined dramatically but COPD is an increasingly recognized but poorly understood complication[14]. A meta-analysis on the epidemiology of COPD in the global HIV-infected population to date demonstrates COPD prevalence between 3 and 23%[15].

Until 2015, the prevalence and risk factors for COPD in Uganda had been largely uncharacterized. The prevalence of COPD was first estimated in a rural population in Uganda at 16% prevalence[11]. In this study, they did not compare prevalence by HIV status. The reported prevalence was higher compared to other studies in the region and may be explained by other factors. Siddharthan and colleagues reported a 6.1% prevalence of COPD in rural Ugandan communities of Nakaseke district compared to a 1.5% prevalence in urban communities of Kampala[16]. In this study, it was highlighted that the most important factor associated with COPD was rural residence, and HIV did not appear to be an important risk factor for COPD[5]. Nevertheless, this population-based study did not explore the effects of HIV viral load and CD4 count on COPD prevalence and lung function outcomes. Also, HIV status was self-reported at 8.1%. Similarly, in a recent study in Southwestern Uganda, North and colleagues did not report any significant association between HIV and respiratory symptoms nor lung function. However, the authors did not explore the effects of HIV-specific characteristics on COPD[17].

In a rural setting of ART clinics in Nakaseke district of Uganda, with participants having well-controlled HIV, we found a COPD prevalence of 6.22%[5]. History of pulmonary tuberculosis was strongly associated with COPD and reduced lung function. As expected, increasing age was associated with reduced lung function. However, HIV specific characteristics including use and duration of ART, current and baseline CD4+T cell counts and viral load were not associated with COPD or reduced lung function both in an adjusted and adjusted analysis[5]. Among those diagnosed, COPD was associated with reduced respiratory health status and severe respiratory symptoms. Currently, it's not fully known what drives chronic lung inflammation in our PLWHA population with over 90% virologically suppressed, cluster of differentiation 4 (CD4) count >500, 80% non-smoker, with history of cure from pulmonary tuberculosis and no significant association between COPD and biomass exposure[5]. Evidence from recent studies suggests that bacterial communities inhabiting mucosal surfaces of airways drive chronic inflammation[8].

Under homeostatic conditions, airway mucosal surface is inhabited by commensal microbial communities. These organisms induce colonization resistance against pathobionts through several molecular mechanisms[18]. The most studied mechanisms involve microbe-microbe and microbe-host interactions. Commensals replicate very rapidly and subsist in densely occupied biological niches, limiting nutrient availability within these micro-habitats. This competition for resources such as amino acids, sugars, zinc, iron and oxygen limits colonization by pathobionts[18]. Thus, a higher microbial diversity implies more microbes utilizing a more versatile pool of metabolites, posing a challenge for any pathobionts to thrive. Therefore, any changes resulting in loss of microbial biomass or diversity destabilizes the microbial ecosystem, creating an opportunity for strains with increased fitness to proliferate.

Some commensals directly inhibit growth of pathobionts through secretion of antimicrobial peptides (AMPs). Such factors restrain the growth of adjacent bacteria by a plethora of mechanisms such as inhibition of cell wall synthesis, formation of pores, and nuclease activity. Other non-peptide molecules that inhibit proliferation of neighboring bacteria include short-chain fatty acids (SCFAs), hydrogen peroxide (H2O2), and secondary bile acids. Finally, bacterial secretion systems (especially Type VI secretion system) have been widely used by commensals to transport toxic substances into their environment or even nearby eukaryotic or prokaryotic cells[18].

ELIGIBILITY:
Inclusion Criteria:

* We will consider samples from Male and female HIV-seropositive and negative individuals ≥35 years who have been screened for COPD as per standard guidelines (European Respiratory Society, ERS, and American Thoracic Society, ATS) using the modified Burden of lung diseases (BOLD) questionnaire and spirometry.

Exclusion Criteria:

* We will exclude samples from subjects with asthma, significant chronic respiratory disease other than COPD or unable to give informed consent.

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected target population:
  80 HIV-infected individuals ≥35 years attending the ART clinic at Nakaseke General Hospital screened for COPD following ERS/ATS guidelines.
  HIV-negative target population:
  80 HIV-negative individuals ≥35 years attending the pulmonary clinic at Nakaseke General Hospital screened for COPD following ERS/ATS guidelines.
  40 stable COPD participants and 40 participants with no COPD exacerbations.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Airway microbial profiling using meta-genomics analysis | Month 12-18
  16S sequencing and metagenomics analysis to determine airway bacterial communities
Airway pro-inflammatory and pro-fibrotic gene expression profiling | Month 12-18
  RNA sequencing and analysis to determine gene expression profiles
Airway immune cellular profiling | Month 12-18
  Airway immune cellular profiling using mass flow time of flight analysis

SECONDARY OUTCOMES:
Role of Out Membrane Vesicles (OMVs) in mediating microbiome effect on airway immune responses | Month 12-18
  ole of Out Membrane Vesicles (OMVs) in mediating microbiome effect on airway immune responses

CONTACTS AND LOCATIONS:
Overall Officials: Alex Kayongo, MD, Principal Investigator — Makerere University Lung Institute
Locations (1):
- Makerere University Lung Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Due to the huge size of the -omics data, access will be through Makerere Lung Institute (MLI) online server, using a fast, secure and optimized data transfer protocol for high-bandwidth networks. The PI will also make copies of meta data available to co-investigators, students, and others by request within 45 days from receipt of the request unless a longer period is necessary for protection of intellectual property after ethical and institutional clearance. We plan to archive and make available by request data that are used to produce published results. We will use email to provide access, depending on the contents of the request. Significant findings from data recorded during the proposed project will be promptly submitted for journal publication. Thus, the most important data will be freely available to all, either as part of journal articles or as supplementary material that is available at the journals' websites.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The PI will also make copies of meta data available to co-investigators, students, and others by request within 45 days from receipt of the request unless a longer period is necessary for protection of intellectual property after ethical and institutional clearance.
  Data will, in principle, be available for access and sharing not later than two years after the acquisition of the data. Key data relevant to the discovery will be preserved until all issues of intellectual property are resolved. Dissemination of data shall be consistent with decisions regarding the management of intellectual property pertaining to the project
Access Criteria: To be determined at a later time

REFERENCES:
- [Background] Stringer JS, Zulu I, Levy J, Stringer EM, Mwango A, Chi BH, Mtonga V, Reid S, Cantrell RA, Bulterys M, Saag MS, Marlink RG, Mwinga A, Ellerbrock TV, Sinkala M. Rapid scale-up of antiretroviral therapy at primary care sites in Zambia: feasibility and early outcomes. JAMA. 2006 Aug 16;296(7):782-93. doi: 10.1001/jama.296.7.782. PMID 16905784
- [Background] Asiki G, Reniers G, Newton R, Baisley K, Nakiyingi-Miiro J, Slaymaker E, Kasamba I, Seeley J, Todd J, Kaleebu P, Kamali A. Adult life expectancy trends in the era of antiretroviral treatment in rural Uganda (1991-2012). AIDS. 2016 Jan 28;30(3):487-93. doi: 10.1097/QAD.0000000000000930. PMID 26765939
- [Background] van Zyl Smit RN, Pai M, Yew WW, Leung CC, Zumla A, Bateman ED, Dheda K. Global lung health: the colliding epidemics of tuberculosis, tobacco smoking, HIV and COPD. Eur Respir J. 2010 Jan;35(1):27-33. doi: 10.1183/09031936.00072909. PMID 20044459
- [Background] Kayongo A, Wosu AC, Naz T, Nassali F, Kalyesubula R, Kirenga B, Wise RA, Siddharthan T, Checkley W. Chronic Obstructive Pulmonary Disease Prevalence and Associated Factors in a Setting of Well-Controlled HIV, A Cross-Sectional Study. COPD. 2020 Jun;17(3):297-305. doi: 10.1080/15412555.2020.1769583. Epub 2020 May 28. PMID 32462945
- [Background] Abt MC, Osborne LC, Monticelli LA, Doering TA, Alenghat T, Sonnenberg GF, Paley MA, Antenus M, Williams KL, Erikson J, Wherry EJ, Artis D. Commensal bacteria calibrate the activation threshold of innate antiviral immunity. Immunity. 2012 Jul 27;37(1):158-70. doi: 10.1016/j.immuni.2012.04.011. Epub 2012 Jun 14. PMID 22705104
- [Background] Le Noci V, Guglielmetti S, Arioli S, Camisaschi C, Bianchi F, Sommariva M, Storti C, Triulzi T, Castelli C, Balsari A, Tagliabue E, Sfondrini L. Modulation of Pulmonary Microbiota by Antibiotic or Probiotic Aerosol Therapy: A Strategy to Promote Immunosurveillance against Lung Metastases. Cell Rep. 2018 Sep 25;24(13):3528-3538. doi: 10.1016/j.celrep.2018.08.090. PMID 30257213
- [Background] Yang D, Chen X, Wang J, Lou Q, Lou Y, Li L, Wang H, Chen J, Wu M, Song X, Qian Y. Dysregulated Lung Commensal Bacteria Drive Interleukin-17B Production to Promote Pulmonary Fibrosis through Their Outer Membrane Vesicles. Immunity. 2019 Mar 19;50(3):692-706.e7. doi: 10.1016/j.immuni.2019.02.001. Epub 2019 Feb 26. PMID 30824326
- [Background] Segal LN, Clemente JC, Tsay JC, Koralov SB, Keller BC, Wu BG, Li Y, Shen N, Ghedin E, Morris A, Diaz P, Huang L, Wikoff WR, Ubeda C, Artacho A, Rom WN, Sterman DH, Collman RG, Blaser MJ, Weiden MD. Enrichment of the lung microbiome with oral taxa is associated with lung inflammation of a Th17 phenotype. Nat Microbiol. 2016 Apr 4;1:16031. doi: 10.1038/nmicrobiol.2016.31. PMID 27572644
- [Background] van Gemert F, Kirenga B, Chavannes N, Kamya M, Luzige S, Musinguzi P, Turyagaruka J, Jones R, Tsiligianni I, Williams S, de Jong C, van der Molen T. Prevalence of chronic obstructive pulmonary disease and associated risk factors in Uganda (FRESH AIR Uganda): a prospective cross-sectional observational study. Lancet Glob Health. 2015 Jan;3(1):e44-51. doi: 10.1016/S2214-109X(14)70337-7. PMID 25539969
- [Background] Celli BR, MacNee W; ATS/ERS Task Force. Standards for the diagnosis and treatment of patients with COPD: a summary of the ATS/ERS position paper. Eur Respir J. 2004 Jun;23(6):932-46. doi: 10.1183/09031936.04.00014304. No abstract available. PMID 15219010
- [Background] GBD 2015 Tobacco Collaborators. Smoking prevalence and attributable disease burden in 195 countries and territories, 1990-2015: a systematic analysis from the Global Burden of Disease Study 2015. Lancet. 2017 May 13;389(10082):1885-1906. doi: 10.1016/S0140-6736(17)30819-X. Epub 2017 Apr 5. PMID 28390697
- [Background] Walker AS, Mulenga V, Ford D, Kabamba D, Sinyinza F, Kankasa C, Chintu C, Gibb DM; CHAP Team. The impact of daily cotrimoxazole prophylaxis and antiretroviral therapy on mortality and hospital admissions in HIV-infected Zambian children. Clin Infect Dis. 2007 May 15;44(10):1361-7. doi: 10.1086/515396. Epub 2007 Apr 12. PMID 17443476
- [Background] Bigna JJ, Kenne AM, Asangbeh SL. Epidemiology of chronic obstructive pulmonary disease in the global HIV-infected population: a systematic review and meta-analysis protocol. Syst Rev. 2017 Mar 29;6(1):68. doi: 10.1186/s13643-017-0467-x. PMID 28356123
- [Background] Siddharthan T, Grigsby M, Morgan B, Kalyesubula R, Wise RA, Kirenga B, Checkley W. Prevalence of chronic respiratory disease in urban and rural Uganda. Bull World Health Organ. 2019 May 1;97(5):318-327. doi: 10.2471/BLT.18.216523. Epub 2019 Mar 26. PMID 31551628
- [Background] North CM, Kakuhikire B, Vorechovska D, Hausammann-Kigozi S, McDonough AQ, Downey J, Christiani DC, Tsai AC, Siedner MJ. Prevalence and correlates of chronic obstructive pulmonary disease and chronic respiratory symptoms in rural southwestern Uganda: a cross-sectional, population-based study. J Glob Health. 2019 Jun;9(1):010434. doi: 10.7189/jogh.09.010434. PMID 31217961
- [Background] Leshem A, Liwinski T, Elinav E. Immune-Microbiota Interplay and Colonization Resistance in Infection. Mol Cell. 2020 May 21;78(4):597-613. doi: 10.1016/j.molcel.2020.03.001. Epub 2020 Mar 23. PMID 32208169
- See also: Organization, W.H., Global status report on noncommunicable diseases 2014. 2014: World Health Organization. — https://apps.who.int/iris/bitstream/handle/10665/148114/9789241564854_eng.pdf
- See also: Organization, W.H., Fact sheet: HIV treatment and care: what's new in HIV treatment. 2015, World Health Organization. — https://apps.who.int/iris/handle/10665/204347